CLINICAL TRIAL: NCT03899272
Title: Positive and Negative Affects Among Osteoarthritis Patient
Brief Title: Psychological Strengths and Burden Among Osteoarthritis Patient
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lawrence CM Lau, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: 2018.113
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee; Psychological
Keywords: osteoarthritis; psychology
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteoarthritis: All new patient present to clinic referred for osteoarthritis for considering joint replacement Present with knee pain (unilateral or bilateral) contributed by osteoarthritis

SUMMARY:
Osteoarthritis (OA) is a common and debilitating disease, For the majority of patients, pain in OA is episodic in nature.

The experience of pain is generated or modified by nociception, neuropathic symptoms, psychological and personality factors, genetic influences, past painful experiences, comorbid conditions, and expectations related to future pain Previous studies have shown psychological well-being has been significantly associated with disability in patients with OA, and anxiety has been found to be associated with knee pain in women.

Previous studies also found that there are large interindividual differences among persons with knee osteoarthritis (OA) with respect to psychological function.

Psychological strengths and weaknesses are evaluated among new patient with osteoarthritis presented to joint replacement clinic, to facilitate our understanding of those patients need, and correlating with their radiological and clinical findings. Psychological strengths and weaknesses, positive and negative affects are evaluated in form of questionaires.

Reference:

Adaptation to disability: Applying selective optimization with compensation to the behaviors of older adults with osteoarthritis.

MAM Gignac, C Cott, EM Badley - Psychology and aging, 2002

Analgesic effects of multisensory illusions in osteoarthritis C Preston, R Newport - Rheumatology, 2011

Psychological factors and their relation to osteoarthritis pain BL Wise, J Niu, Y Zhang, N Wang, JM Jordan… - Osteoarthritis Cartilage. , 2010 - Elsevier

DETAILED DESCRIPTION:
Introduction:

Osteoarthritis (OA) is a prevalent painful condition that may cause disability among older adults (Cruz-Almeida et al., 2013). Psychological traits and emotional states of patients were found to be correlated with symptoms of OA and daily functioning of patients (Cruz-Almeida et al., 2013; Dezutter et al., 2015).

The experience of pain is generated or modified by nociception, neuropathic symptoms, psychological and personality factors, genetic influences, past painful experiences, comorbid conditions, and expectations related to future pain. Previous studies have shown psychological well-being has been significantly associated with disability in patients with OA, and anxiety has been found to be associated with knee pain in women.

Previous studies also found that there are large interindividual differences among persons with knee osteoarthritis (OA) with respect to psychological function.

Aim of project:

This research is trying to find out what psychological strengths or factors could attenuate the chronic pain of knee OA patients. The purpose of the study is to find psychological evidences that may be used in the future to help chronic pain patients for improving their daily functioning and well-being.

ELIGIBILITY:
Inclusion Criteria:

* all new patient present to AHNH clinic referred for osteoarthritis for considering joint replacement
* Present with knee pain (unilateral or bilateral) contributed by osteoarthritis

Exclusion Criteria:

* mentally unsound
* dialectic speaker that difficult to communicate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 150 patients, based on previous studies (Psychological Proﬁles and Pain Characteristics of Older Adults With Knee Osteoarthritis; Psychological factors and their relation to osteoarthritis pain) and the number of patients and study time available in our clinic
  Those are all the new patient present to AHNH clinic referred for osteoarthritis for considering joint replacement
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Scale (PANAS) | 1 day
  This scale consists of a number of questions that describe different feelings and emotions.
The Centre for Epidemiologic Studies (CES-D Scale) | 1 day
  A list of the ways the subject might have felt or behaved.
The Chronic Pain Acceptance Questionnaire (CPAQ) | 1 day
  Statements on feelings on pain as it applies to the subject.
Chronic Pain Coping Inventory (CPCI-42) | 1 day
VIA-72 | 1 day
  Questions reflect statements that the subject would find desirable.
Kellgren & Lawrence (K & L) grading system | 1 day
  To classify the severity of knee osteoarthritis (OA)
Oxford knee scores | 1 day
  Consists of 12 questions that cover function and pain of the knee.

CONTACTS AND LOCATIONS:
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: No